CLINICAL TRIAL: NCT02523703
Title: Excitotoxicity Markers and the Clinical-radiological Progression After a Demyelinating Event: a Prospective Pilot Study
Acronym: EXCEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 06-063
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Glutamic Acid; Aspartic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Other): Healthy Volunteers
  Interventions: Biological: glutamate and aspartate
- Multiple Sclerosis patient (Other): Multiple Sclerosis patient
  Interventions: Biological: glutamate and aspartate

INTERVENTIONS:
Biological: glutamate and aspartate

SUMMARY:
Multiple sclerosis (MS) is an inflammatory disease of the central nervous system, beginning most often in subjects aged 20-40 years. In France, thanks to recent studies reported during general states of MS in 2006, the prevalence is estimated at 65.5 / 100,000 population (96.3 / 100,000 women and 41.9 / 100,000 men) and incidence at 7.91 per 100,000. In Lower Normandy, the incidence of MS is estimated to 4.45 / 100,000 inhabitants or 60 new cases per year.

The primary objective of this pilot study is to assess the levels of glutamate and aspartate (excitotoxicity markers) and their repercussions on the clinical and radiological outcome in 40 patients experiencing an event demyelinating central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 and 60 years old.
* Patient with one or more type of inflammatory events of Central system suggestive of demyelinating disease (multiple sclerosis, neuromyelitis optical Devic extensive myelitis)
* No treatment with corticosteroids for less than 1 month
* Need for a lumbar puncture performed in the etiologic
* Need a brain MRI performed within the etiologic
* Patient who signed informed consent

Exclusion Criteria:

* Secondary progressive MS
* Any cons-indication for lumbar puncture
* Any contra-indication to MRI
* Minor patient or patient major under guardianship

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-09-10 (Actual); Primary Completion 2012-02-15 (Actual); Study Completion 2015-02-23 (Actual)

PRIMARY OUTCOMES:
glutamate concentration (in nM) | baseline
  comparison between MS patients and controls